CLINICAL TRIAL: NCT00400244
Title: Translation, Validation and Evaluation of the Efficacy of the French-Canadian Version of the Wheelchair Skills Program (WSP)
Brief Title: French-Canadian Version of the Wheelchair Skills Program (WSP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: François Routhier, CIRRIS
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA009
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-01

CONDITIONS: Disabled Persons
Keywords: wheelchairs; skills; french

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Wheelchair skills traing program

SUMMARY:
The purpose of this project is to develop French Canadian versions of the Wheelchair Skills Program (WSP). Translating a measurement instrument in the field of biomedical sciences requires not only the language to be taken into account but also the cultural context. We will determine the measurement properties of the WST-F and complete the randomized controlled trial on the efficacy of the WSTP-F.

ELIGIBILITY:
Inclusion Criteria:

* eighteen (18) or older;
* use a manual wheelchair at least four (4) hours per day;
* in the rehabilitation process (including training in manual wheelchair use);
* have enough ability to develop skills included in the wheelchair skills training program;
* are willing to take part in the study;
* French-speaking individual capable of understanding enough of the English language to sign this form after carefully reading it
* competent to give informed consent or have a proxy with power of attorney;
* have the verbal endorsement of the clinical therapist (if any) to participate;
* have the permission of the attending physician or occupational therapist to participate;
* are alert and cooperative.

Exclusion Criteria:

* have an unstable medical condition (e.g. angina, seizures), as indicated by the attending physician, hospital or rehabilitation centre staff, enhanced registered nurse or self-report;
* have an emotional or psychiatric problem of a type or extent that might make participation unpleasant, as indicated by the attending physician, hospital or rehabilitation centre staff, enhanced registered nurse or self-report.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
French version of the Wheelchair Skills Test

CONTACTS AND LOCATIONS:
Overall Officials: Francois Routhier, PhD, Principal Investigator — Institut universitaire de geriatrie de Montreal
Locations (1):
- Centre de recherche interdisciplinaire en readaption, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Routhier F, Kirby RL, Demers L, Depa M, Thompson K. Efficacy and retention of the French-Canadian version of the wheelchair skills training program for manual wheelchair users: a randomized controlled trial. Arch Phys Med Rehabil. 2012 Jun;93(6):940-8. doi: 10.1016/j.apmr.2012.01.017. Epub 2012 Apr 10. PMID 22494946